CLINICAL TRIAL: NCT06034288
Title: IncobotulinumtoxinA (Xeomin®) vs OnabotulimuntoxinA (Botox®) for Treatment of Overactive Bladder Syndrome: Randomized Non-Inferiority Trial
Brief Title: Xeomin vs Botox for Treatment of Overactive Bladder Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WRNMMC-2022-0398
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Xeomin (Experimental): 100units xeomin dilated in 10mL injectable saline will be injected into the detrusor muscle to a depth of 3mm at 20 sites at 0.5mL volume each
  Interventions: Drug: Xeomin 100 UNT Injection
- Botox (Active Comparator): 100units Botox dilated in 10mL injectable saline will be injected into the detrusor muscle to a depth of 3mm at 20 sites at 0.5mL volume each
  Interventions: Drug: Botox 100 UNT Injection

INTERVENTIONS:
Drug: Xeomin 100 UNT Injection — intravesical injection
  Other Names: incobotulinumtoxinA
  Arms: Xeomin
Drug: Botox 100 UNT Injection — intravesical injection
  Other Names: onabotulinumtoxinA
  Arms: Botox

SUMMARY:
Purpose: Multiple formulations and brands of botulinum toxin exist on the market today. Only OnabotulinumtoxinA (BOTOX®) is currently FDA approved for treatment of overactive bladder. IncobotulinumtoxinA (XEOMIN®) is a similar formulation of botulinum toxin A that has similar dosing and safety profile at onabotulinumtoxinA. OnabotulinumtoxinA is the most expensive formulation on the market. Compare the efficacy of incobotulinumtoxinA (Xeomin®, Merz Pharmaceuticals) to onabotulinumtoxinA (Botox®, Allergan) for treatment of OAB. Study design: A single-blinded, randomized non-inferiority trial of IncobotulinumtoxinA (Xeomin®, Merz Pharmaceuticals) to OnabotulinumtoxinA (Botox®, Allergan) in treatment of OAB. Target Population: The study findings will be applicable to all women 18 years of age or older with OAB symptoms associated with urinary urgency incontinence. Procedure: All patients that presents to urogynecology clinic at Walter Reed National Medical Military Center will be screened for inclusion and exclusion criteria. Patients that meet criteria will be offered to participate in the study. After enrollment patient will complete demographics data sheet, 24 hours bladder diary, OAB-q SF, PGI-S, PISQ-IR. Patients will be randomized by the principal investigator and the allocated treatment will be reveled by the treating provider to the treating provider only. Patient will have a follow up at 2-6 weeks and 6-9 months after procedure. During the follow up appointments patient will be asked to fill out 24-hour voiding diary, OAB-q SF, PGI-I, PGI-S, and PISQ-IR surveys.

DETAILED DESCRIPTION:
The study will be registered on clinicaltrials.gov after IRB approval. Institutional Review Board (IRB) approval will be received.

All women 18 years of age and older with bothersome overactive bladder symptoms who are receiving care at Walter Reed National Military Medical Center (WRNMMC) in the urogynecology clinic will be eligible for the study.

All study participants will undergo a complete intake assessment to include a history, physical exam, post-void bladder residual volume assessment via straight catheterization or ultrasound, and counseling on treatment modalities for OAB using the AUGS handout to include behavioral and dietary modifications, physical therapy, oral medications, onabotulinumtoxinA and neuromodulation. Patients desiring treatment with onabotulinumtoxinA will be scheduled for the procedure. Patients do not have to fail prior treatment options in order to qualify for bladder BOTOX. This is all standard of care in our practice. All patients meeting the inclusion and exclusion criteria will be offered enrollment in this study. Enrollment will be done by the research team, who typically are also the clinicians. No patients will be pressured or coerced into participating in the study.

Prior to the procedure appointment, participants will be consented for participation in the study and asked to complete demographics data sheet, 24 hours bladder diary, OAB-q SF, PGI-S, PISQ-IR. OAB-q SF is a standard of are in our practice, all other questionnaires patient will fill out for the purpose of this study.

The procedure will be performed at Walter Reed National Military Medical Center either in clinic setting or in the operating room. All patients who plan to undergo the procedure in clinic will be offered a pre-treatment anxiolytic with a single dose of 5-10mg of oral diazepam, which is standard practice at this institution. Patients undergoing the procedure in the operating room, will be given sedation medications as per standard of care. As standard of treatment, patients will also be given a prescription for an antibiotic - either nitrofurantoin 100mg to take orally twice daily for 3 days starting the day of the procedure, or trimethoprim-sulfamethoxazole 800mg-160mg to take orally twice daily for 3 days starting the day of the procedure depending on patient's allergy profile.

The principal investigator will make randomized assignments using the RAND function in excel. The first 32 random numbers will be assigned to BOTOX arm and the second 32 numbers will be assigned to XEOMIN arm. Each assignment number will be placed in a sealed envelop by the PI. The sealed envelops will be opened by the treatment provider the day of the scheduled procedure. The envelop will reveal the medication assignment to the provider. After the provider reveals the medication only to him/herself (not the patient), the appropriate medication will be obtained from the pharmacy and administered to the patient.

The patient will be blinded to the treatment allocation. The drug will be obtained from the pharmacy on the day of the procedure by the treatment team. Either onabotulinumtoxinA or incobotulinumtoxinA (as determined by the allocated assignment), will be reconstituted in 10 milliliters of injectable saline by the treatment team prior to entering the patient's room, to keep the patient blinded. The bladder will be filled with 20ml of 2% viscous lidocaine through the urethra 15 to 20 minutes prior to the procedure per the Urogynecology department standard operating procedure for intradetrusor onabotulinumtoxinA injections. Operative cystoscopy will be performed, and an adjustable-depth injection cystoscopy needle will be used to inject the blinded study drug (either 100 units of onabotulinumtoxinA (Botox®, Allergan) or 100 units of incobotulinumtoxinA (Xeomin®, Merz Pharmaceutical)) with the needle depth set to 3mm. Injections will be performed by either a board-certified staff Urogynecologist, or fellows or residents working under their direct supervision of the board-certified staff urogynecologist. An injection cystoscopy needle will be set to 3mm and used to inject 0.5mL reconstituted study medication at each injection site, approximately 1cm apart along the posterior bladder wall making sure to avoid the trigone, for a total or 20 injection sites (4 rows of 5 injection sites). After the completion of the procedure, patients will be asked to start taking their prescribed antibiotics and to continue them for 3 days.

If a known UTI was inadequately treated prior to procedure appointment, or if there is evidence of an active infection at the time of cystoscopy, the intravesical injection will not be completed and patient will be rescheduled.

Participants will have a follow-up appointment in 2-6 weeks following the procedure in person, via phone or email. At the follow-up visit patients will be asked to complete a 24-hour bladder diary, OAB-q SF, PGI-I, PGI-S, PISQ-IR surveys. The surveys will either be read or emailed to the patient based on patient's preference. Patients will be asked regarding urinary tract infection (UTI) symptoms and whether they needed clean intermittent catheterization (CIC). The electronic health record (EHR) will also be reviewed to confirm whether UTI has occurred or if CIC needed to be done. Patients will be asked whether they are experiencing painful urination, urinary frequency, urinary urgency, or blood in their urine. If patients answer yes to any of those questions, they will be asked to provide a urine sample. If this follow up is being done in person, then a urine sample will be obtained via straight catheterization during the appointment. If the follow up visit is being done virtually, patient will be asked to come into clinic or laboratory and provide a urine sample via straight catheterization or clean catch for urinalysis and urine culture to assess for UTI. If infection is present, patients will receive appropriate antibiotics based on culture sensitivities. Patients found to have an active infection at the time of postprocedural follow-up will be asked to complete the study questionnaires 2-4 weeks following treatment of infection. Patients will also be asked if they experienced any other symptoms following the procedure that concerned them and any symptoms reported will be recorded.

Participants who experience initial relief in their symptoms following injection of the study medication but then experience recurrence of symptoms will be eligible for repeat injection provided it has been at least 12 weeks from prior injection and the total dose of onabotulinumtoxinA/incobotulinumtoxinA does not exceed 400 units in a three-month time frame, as is standard of care.

Six to nine months following the treatment, patients will be contacted via phone or email and asked to complete a 24-hour voiding diary, OAB-q SF, PGI-I, PGI-S, and PISQ-IR surveys for final assessment of symptoms following treatment. They will again be asked regarding adverse events. The questionnaires again will either be read to the patient via phone or emailed based on patient's preference.

This research study is a single-blind study. Unblinding of subjects will be performed at the conclusion of the study after enrollment is closed and data collection is complete. Participants will not be notified of their group assignment unless it is requested after the completion of the final follow up encounter. If the participant would like to know their group assignment, they will contact the PI who will release that information to them after the conclusion of the study. Study participants who request to be un-blinded as to their randomized assigned group early will need to be withdrawn from the study. The participant will supply a request in writing to the PI. Any data regarding that participant will be removed from the records and that assignment number will be noted as withdrawn. A memorandum for record will be created outlining the subject's request and both the MFR and subject's written request will be maintained with the data collection for reference. In the event of an emergency, there is a way to find out which one the participant is receiving. If there is a medical emergency that may require unblinding prior to the conclusion of the study, the research team will work in coordination with the subject's primary care or emergency provider to determine if unblinding is necessary and make that information available to them as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years of age or older
2. Primary complaint of urinary urgency incontinence
3. Failed at least one medication (inadequate or poorly tolerated response) or behavior modification technique (timed voiding, pelvic floor physical therapy, dietary modifications, etc.), or decline such interventions
4. Willingness to perform self-catheterization
5. Ability to follow study instructions and complete all required follow-up
6. DEERS eligible

Exclusion Criteria:

1. Concurrent use of oral medications for treatment of OAB (anticholinergics or beta 3 agonists)
2. Contraindication to onabotulinumtoxinA and/or incobotulinumtoxin
3. Post void residual volume > 200 ml
4. Symptomatic prolapse POP-Q (Pelvic Organ Prolapse Quantification) stage three or greater that is untreated
5. Evidence of active bladder infection
6. Any previous use of intradetrusor botulinum toxin within the preceding 6 months
7. Total body onabotulinumtoxinA and/or incobotulinumtoxinA dose of ≥ 400 Units in the 3 months prior to scheduled appointment
8. Procedure performed in the main operating room (not outpatient setting)
9. Concurrent diagnosis of interstitial cystitis/painful bladder syndrome
10. Females who are pregnant or planning a pregnancy during the study or who think that they may be pregnant at the start of the study, or females of childbearing potential who are unable or unwilling to use a reliable form of contraception during the study
11. Neurogenic bladder or other neurological disease that may cause voiding dysfunction
12. Inability to speak or read English. Non-English speakers will be excluded from this study for ease of being able to allow the principal investigator to communicate with the patients during the consents, initial and all follow-up communication. Some of the questionnaires used have also only been validated in English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Urge urinary incontinence episodes | 2-6 weeks
  To evaluate non-inferiority of incobotulinumtoxinA to onabotulinumtoxinA for treatment of OAB by using number of incontinence episodes on a 24-hours bladder diary at 2-6 weeks post injection

CONTACTS AND LOCATIONS:
Overall Officials: Anna S Trikhacheva, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No